CLINICAL TRIAL: NCT00400556
Title: A Phase I Study of Haematopoietic Stem Cell Mobilization Using G-CSF With ATRA in Patients With Cutaneous Lymphoma and Multiple Myeloma
Brief Title: ATRA Plus G-CSF for Mobilization of Hematopoietic Stem and Progenitor Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04/24
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2006-11-17 (Estimated); Status verified 2006-11

CONDITIONS: Multiple Myeloma; Cutaneous Lymphoma
Keywords: mobilization; ATRA; G-CSF; filgrastim; retinoids; stem cell mobilization; hematopoietic stem and progenitor cells
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, T-Cell, Cutaneous | interventions — Tretinoin; Granulocyte Colony-Stimulating Factor; Filgrastim

INTERVENTIONS:
Drug: ATRA plus G-CSF (filgrastim, NEUPOGEN (R)) combination

SUMMARY:
Hematopoietic stem and progenitor cells (HSPC) are used for transplantation in patients undergoing high dose therapy for the treatment of a range of cancers.

* HSPC are collected from the bloodstream after treatment with medications that cause the HSPC to move from the bone marrow into the bloodstream, a process called mobilization
* between 5 and 60% of patients can fail to collect enough HSPC for a transplant, using current mobilization techniques
* this study aims to assess the safety of combining a derivative of vitamin A, ATRA with G-CSF (the drug most commonly used to mobilize HSPC)
* ATRA has never been combined with G-CSF for mobilization of HSPC and therefore a study is needed to assess the safety of this combination, and whether it successfully mobilizes HSPC

DETAILED DESCRIPTION:
HSPC mobilization is normally achieved using cytokines such as G-CSF, or occasionally GM-CSF, often in combination with myelosuppressive chemotherapy.

Studies in the mouse model have shown that retinoids (vitamin A derivatives) can be combined with G-CSF, and that this combination synergizes to enhance HSPC mobilization over that seen with G-CSF alone.

This trial aims to assess the safety and mobilization efficacy of combining mobilizing doses of G-CSF with a standard dose of ATRA, using a treatment regimen derived from the earlier murine studies.

In this phase I pilot study, six patients with multiple myeloma or cutaneous lymphoma will be treated with ATRA plus G-CSF, and safety and toxicity data collected for the two week study drug period plus a further two weeks' follow-up. The primary endpoint is safety and toxicity, the secondary endpoint is an observation of the mobilization efficacy as demonstrated by CD34+ cell counts over the study period. Patients will not undergo stem cell collection during this study, as this is purely an observational study. Participating patients will not be those who would normally be scheduled for stem cell collection and transplantation in the near future, but rather patients with stable disease who are not candidates for imminent transplantation, or who have collected adequate HSPC on previous mobilization attempts and are currently being observed.

Cutaneous lymphoma and multiple myeloma are chosen as suitable disease states for this study as there is in vitro evidence of a possible disease benefit of retinoids in these disorders. If disease response is noted during the study or follow up period, ongoing ATRA will be offered at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* likely to comply with study protocol
* age of 18-70
* histologically proven multiple myeloma or lymphoma
* not currently receiving cytotoxic agents however thalidomide, prednisolone, dexamethasone are allowable
* multiple myeloma patients must be receiving regular bisphosphonates
* absolute neutrophil count between 1.5 and 10.0 x 10^9/L
* ECOG performance status </= 3
* life expectancy of at least two months
* written informed consent signed by patient or legally authorised representative

Exclusion Criteria:

* use of other vitamin A preparations within the last 30 days
* active infection or fever >/= 38.2 degrees celsius
* pregnancy or breast feeding. Women of child bearing potential admitted to the trial must take adequate measures to prevent conception (at least two different forms of contraception) and are to undergo a pregnancy test. Oral contraception must not include low-dose progestogens
* known allergy to E.coli derived products
* current treatment with tetracycline antibiotics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6
Dates: Start 2005-03; Study Completion 2005-05

PRIMARY OUTCOMES:
Toxicity data (NCI-CTC version 2.0 criteria)
skin toxicity
hepatotoxicity
mucosal toxicity
hematologic toxicity
neurologic toxicity
treatment response
CD34+ cell count peak level
time to CD34+ count peak level
time to reach level >5 x 10^6.L
area under curve for duration of time spent with CD34+ count >5 x 10^6/L
peripheral blood colony forming unit assays
peak CFU-GEMM level
time to peak CFU-GEMM level

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten E Herbert, MBBS, Principal Investigator — Peter MacCallum Cancer Center; Miles Prince, MBBS, Principal Investigator — Peter MacCallum Cancer Center
Locations (1):
- Peter MacCallum Cancer Center, East Melbourne, Victoria, Australia

REFERENCES:
- [Background] Herbert KE, Walkley CR, Winkler IG, Hendy J, Olsen GH, Yuan YD, Chandraratna RA, Prince HM, Levesque JP, Purton LE. Granulocyte colony-stimulating factor and an RARalpha specific agonist, VTP195183, synergize to enhance the mobilization of hematopoietic progenitor cells. Transplantation. 2007 Feb 27;83(4):375-84. doi: 10.1097/01.tp.0000251376.75347.b4. PMID 17318068